CLINICAL TRIAL: NCT00169481
Title: A Randomized, Controlled, Phase II Study to Evaluate the Safety and Immunogenicity of Different Formulations of GlaxoSmithKline Biologicals' 11-valent Pneumococcal Conjugate Vaccine, When Administered Intramuscularly as a 3-dose Primary Immunization (2-3-4 Month Schedule) Before 6 Months of Age
Brief Title: A Study in Children With Different Formulations of GSK Biologicals' 11 Valent Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 103488
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Streptococcal Infections
MeSH Terms: conditions — Streptococcal Infections | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Biological: Pneumococcal (vaccine)

SUMMARY:
Three dose primary vaccination with 11-valent pneumococcal conjugate vaccine administered concomitantly with Infanrix™ hexa to healthy infants between 8 to 16 weeks of age at the time of first vaccination.

DETAILED DESCRIPTION:
Test groups: 9 groups receiving different formulations of 11PN-PD-DiT vaccine + DTPa-HBV-IPV/Hib (Infanrix™ hexa) Comparator: 11Pn-PD + Infanrix™ hexa Control: Prevenar® + Infanrix™ hexa

ELIGIBILITY:
Inclusion criteria:

* Male or female aged 8-16 weeks at the time of first vaccination, written informed consent obtained from the parent/guardian of subject.

Exclusion criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceeding the first dose of study vaccine, or planned use during the study period.
* Planned administration/ administration of a licensed vaccine not foreseen by the study protocol during the period starting from 30 days before the first dose of vaccine(s) and ending 30 days after the last dose.

Ages: 8 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 689 (Actual)
Dates: Start 2004-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
1 month after d3, antibody concentrations to pneumo. serotypes 1,3,4,5,6B,7F,9V,14,18C,19Fand23F.Occurrence of: solicited local and general symptoms within 8 days after each vaccination; unsolicited adverse events within 31 days after each vaccination | 1 Month after dose 3

SECONDARY OUTCOMES:
1 month post d3: For pneumo.serotypes 1,3,4,5,6B,7F, 9V,14,18C,19F,23F:Opsono titres;antibody concentrations (AbC) >= 0.20 µg/mL;AbC to protein D and seropositivity (S+)status; S+/seroprotection status to antigens in Infanrix hexa. | 1 Month after dose 3

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- Germany (48):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bretten, Baden-Wurttemberg
  - GSK Investigational Site, Eppelheim, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Herzogenaurach, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Zwiesel, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Koenigstein, Hesse
  - GSK Investigational Site, Marburg/Lahn, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Waren, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Bodenheim, Rhineland-Palatinate
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Schoeneberg - Kuebelberg, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Bredstedt, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Neumünster, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Weimar, Thuringia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 103488 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103488 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103488 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103488 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103488 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register